CLINICAL TRIAL: NCT00884325
Title: Management of Pruritus With Xyzal in Atopic Dermatitis in a Randomized, Double-Blind, Placebo Controlled Study
Brief Title: Management of Pruritus With Xyzal in Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Leon Kircik, M.D., Principal Investigator, Derm Research, PLLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XYZ0801
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Results first posted 2013-08-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Atopic Dermatitis; Pruritus
Keywords: Itching; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xyzal (Experimental)
  Interventions: Drug: Levocetirizine dihydrochloride (Xyzal)
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Levocetirizine dihydrochloride (Xyzal) — One tablet 5 mg taken orally at night for 28 days
  Other Names: Xyzal
  Arms: Xyzal
Drug: placebo — One tablet taken orally at night for 28 days
  Arms: Placebo

SUMMARY:
It is historically well known that the management of pruritus in atopic dermatitis is very difficult. Most of the patients are not controlled with traditional antihistamines such as Clarinex, Claritin, and Allegra. It will be a welcome addition to our treatment armamentarium if a drug such as Xyzal can control pruritus associated with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female subjects of any race, at least 18 years of age.
* Female subjects of childbearing potential must have a negative urine pregnancy test result at Baseline and practice a reliable method of contraception throughout the study. A female is considered of childbearing potential unless she is:

  * postmenopausal for at least 12 months prior to study drug administration;
  * without a uterus and/or both ovaries; or
  * has been surgically sterile for at least 6 months prior to study drug administration.
* Reliable methods of contraception are:

  * hormonal methods or intrauterine device in use > 90 days prior to study drug administration;
  * barrier methods plus spermicide in use at least 14 days prior to study drug administration; or
  * vasectomized partner. [Exception: Female subjects of childbearing potential who are not sexually active will not be required to practice a reliable method of contraception. These subjects may be enrolled at the Investigator's discretion if they are counseled to remain sexually inactive during the study and understand the possible risks in getting pregnant during the study.]
* Definitive diagnosis of atopic dermatitis as per Rajka-Hanifin criteria.
* Visual Analog Scale (VAS) pruritus score of 6 cm or more (moderate to severe itching) at baseline.
* Willing to refrain from other antihistamines and topical steroids and topical immunomodulators for the duration of the study.
* Able to understand and comply with the requirements of the study and sign Informed Consent/Health Insurance and Portability Accountability Act (HIPAA) Authorization forms.

Exclusion Criteria:

* Female subjects who are pregnant (positive urine pregnancy test), breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
* Requiring oral treatment for their atopic dermatitis apart from oral antihistamines
* History of hypersensitivity or idiosyncratic reaction to to any component of the test medication , or to cetirizine.
* Atopic Dermatitis triggered by an unavoidable irritant/allergen.
* Skin disease/disorder that might interfere with the diagnosis or evaluation of atopic dermatitis (e.g., erythroderma, skin infection on the affected area, etc.)
* Non-compliance with the proper wash-out periods for prohibited medications.
* Uncontrolled chronic disease such as diabetes
* The presence of renal disease with mild, moderate or severe renal impairment
* Medical condition that, in the opinion of the Investigator, contraindicates the subject's participation in the clinical study.
* Clinically significant alcohol or drug abuse, in the opinion of the Investigator.
* History of poor cooperation, non-compliance with medical treatment, or unreliability.
* Participation in an investigational drug study within 30 days of the Baseline Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon H. Kircik, M.D., Principal Investigator — DermResearch, PLLC
Locations (1):
- DermResearch, PLLC, Louisville, Kentucky, United States

REFERENCES:
- [Background] Hannuksela M, Kalimo K, Lammintausta K, Mattila T, Turjanmaa K, Varjonen E, Coulie PJ. Dose ranging study: cetirizine in the treatment of atopic dermatitis in adults. Ann Allergy. 1993 Feb;70(2):127-33. PMID 8430920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with uncomplicated atopic dermatitis were recruited form the PI's medical practice. Recruitment occurred from March 2009 through December 2009.
Pre-assignment Details: 45 subjects were consented but 5 were screen failures.
Groups:
- Subjects Receiving Xyzal: one tablet, 5 mg, taken orally at night for 28 days
- Subjects Receiving Placebo: one tablet taken orally at night for 28 days
Period: Overall Study
Arm/Group | Subjects Receiving Xyzal | Subjects Receiving Placebo
Started | 20 | 20
Completed | 17 | 16
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Not provided | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects Receiving Xyzal | Subjects Receiving Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age Categorical [Number; unit: participants] — Age data was unknown for one placebo participant
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 19 | 18 | 37
    >=65 years | 1 | 1 | 2
Age Continuous [Mean (Full Range); unit: years] — Age data was missing for one placebo participant
  years | 41.1 (14.6) [19.5 to 64.6] | 41.1 (14.8) [19.8 to 68.1] | 41.1 (14.6) [19.5 to 68.1]
Gender [Number; unit: participants] — gender data was missing for one participant
  participants
    Female | 14 | 12 | 26
    Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Pruritus VAS Scores at Baseline, Week 2 and Week 4
Description: Consented subjects who met inclusion/exclusion criteria were assigned either 5mg levocetirizine dihydrochloride (Xyzal) or placebo to be taken daily each evening for 28 days. Subjects were asked to complete a Visual Analog Scale to measure itch at Baseline, Week 2 and Week 4. The scale is an eleven point scale ranging from 0-10 with 0 indicating no itch to 10 indicating itch that frequently interferes with daily activities.
Time Frame: Baseline - Week 2-Week 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Subjects Receiving Xyzal | Subjects Receiving Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 7.8 [6.5 to 8.5] | 7.5 [7.00 to 8.00]
  Week 2 | 6.10 [1.6 to 7.5] | 5.9 [3.65 to 7.75]
  Week 4 | 4.15 [2.4 to 6.9] | 6.4 [2.5 to 7.3]

2. Secondary Outcome: Dermatology Life Quality Index (DLQI) Questionnaire Scores at Baseline, Week 2 and Week 4
Description: Consented subjects who met inclusion/exclusion criteria were asked to complete a DLQI (Dermatology Life Quality Index)at Baseline, Week 2 and Week 4. The DLQI is a 10 item questionnaire broken down into 6 domains; symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment with a total score ranging from 0-30 (no effect on subject's life for 0, extremely large effect on subject's life for 30)
Time Frame: Baseline - Week 2 - Week 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Subjects Receiving Xyzal | Subjects Receiving Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  DLQI - Baseline | 7.5 [4.00 to 14.00] | 8.00 [7.00 to 13.00]
  DLQI - Week 2 | 3.5 [2.00 to 6.5] | 5.5 [2.00 to 9.00]
  DLQI - Week 4 | 2.00 [1.00 to 5.00] | 4.00 [1.00 to 7.5]

ADVERSE EVENTS:
Arm/Group | Subjects Receiving Xyzal | Subjects Receiving Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 4/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Receiving Xyzal (N=20) | Subjects Receiving Placebo (N=20)
pruritus - worsening (General disorders) | 2 (2) | 1 (1)
seasonal allergies - worsening (Immune system disorders) | 1 (1) | 1 (1)
sinus infection (Infections and infestations) | 1 (1) | 1 (1)
headache (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of subjects. Of 40 subjects enrolled, only 33 completed the 4 week study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No